CLINICAL TRIAL: NCT06123806
Title: Factors Affecting Dialysis Associated Fatigue
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Eldin Hassan Aly Sayed, Candidate of master degree in nephrology, Assiut University
Other Study IDs: dialysis associated fatigue
Record Dates: First submitted 2023-09-23; First posted 2023-11-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dialysis; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the factors affecting hemodialysis-associated fatigue and their impact on the physical and emotional well-being of patients. By identifying these factors, Investigators can develop effective strategies to reduce fatigue and enhance the overall quality of life for hemodialysis patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a significant public health issue affecting millions of individuals worldwide. Hemodialysis, the most common modality for renal replacement therapy, is a life-sustaining procedure for end-stage renal disease (ESRD) patients. Despite its benefits, hemodialysis can be associated with various complications, and one of the most commonly reported symptoms is fatigue. Hemodialysis-associated fatigue (HAF) is characterized by persistent tiredness, lack of energy, and reduced motivation, which significantly impacts the quality of life and functional capacity of patients.

Several potential factors contribute to HAF, including patient-related variables, dialysis-related factors, and comorbidities. Understanding the underlying mechanisms and factors contributing to HAF is essential for improving the overall care and quality of life of hemodialysis patients. Targeted interventions to address fatigue could lead to better adherence to dialysis treatment, reduced hospitalizations, and enhanced overall well-being for this vulnerable patient population. To date, limited research has been conducted on the subject of HAF, and the available studies often have small sample sizes and diverse methodologies. Therefore, this research aims to delve into the complexities of HAF, exploring its prevalence, potential risk factors, and implications for patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult hemodialysis patients aged ≥ 18 years
* patients on hemodialysis for at least 3 months

Exclusion Criteria:

* patients aged < 18 years
* patients with acute kidney injury
* patients with cognitive impairment or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenient sample of adult hemodialysis patients (age ≥ 18 years) who have been on hemodialysis for at least 3 months will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Factors affecting dialysis associated fatigue | baseline
  The aim of this study is to investigate the factors affecting hemodialysis-associated fatigue and their impact on the physical and emotional well-being of patients.

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21993585/
- See also: Related Info — https://www.nature.com/articles/s41581-020-0268-7
- See also: Related Info — https://www.gehealthcare.com/products/contrast-media/visipaque?utm_campaign=PDx-US-22-October-Visipaque-PaidSearch&utm_source=google&utm_medium=cpc&utm_content=website&utm_term=kidney
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31582227/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17345690/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11114998/